CLINICAL TRIAL: NCT04771351
Title: A Randomized, Blinded-controlled Study to Evaluate the Safety and Efficacy of a Single Dose of STI-2020 (COVI-AMG™) in Hospitalized Adult Patients With COVID-19
Brief Title: Study to Evaluate a Single Dose of STI-2020 (COVI-AMG™) in Hospitalized Adults With COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A different study will be conducted.
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMG-COV-202
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Covid19
Keywords: covid-19
MeSH Terms: conditions — COVID-19 | interventions — STI-2020

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- COVI-AMG 100 mg (Experimental): A single injection of 100 mg of COVI-AMG will be administered.
  Interventions: Biological: COVI-AMG
- COVI-AMG 200 mg (Experimental): A single injection of 200 mg of COVI-AMG will be administered.
  Interventions: Biological: COVI-AMG
- Placebo (Placebo Comparator): A single injection of placebo will be administered.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: COVI-AMG — COVI-AMG is a fully human SARS-CoV-2 neutralizing monoclonal antibody (mAb)
  Other Names: STI-2020
  Arms: COVI-AMG 100 mg; COVI-AMG 200 mg
Drug: Placebo — Diluent solution
  Arms: Placebo

SUMMARY:
This is a placebo-controlled study to investigate the safety and efficacy of a single injection of COVI-AMG in inpatient adults with COVID-19.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study designed to investigate the safety and efficacy of a single injection of COVI-AMG in inpatient adults with COVID-19. Subjects will receive 100 mg of COVI-AMG, 200 mg of COVI-AMG, or placebo via slow IV push. Subjects will be followed for approximately 70 days post dosing.

ELIGIBILITY:
Inclusion Criteria:

* Positive for COVID-19 by an approved antigen test
* Progressive disease suggestive of ongoing COVID-19 infection
* Requires hospitalization for acute medical care
* Provides written informed consent
* Willing to follow contraception guidelines during study

Exclusion Criteria:

* Requires high-flow oxygen supplementation
* Current or imminent respiratory failure
* Has rapidly progressing symptoms that in the investigator's opinion are likely to progress to needing high-flow oxygen or to respiratory failure within 24 to 48 hours
* Any condition which, in the investigator's opinion, participation would not be in the subject's best interest or could prevent, limit, or confound the protocol-specified assessments
* Has participated, or is participating in, a clinical research study evaluating COVID-19 convalescent plasma, monoclonal antibodies against SARS-CoV-2, or intravenous immunoglobulin within 3 months or less than 5 half-lives of the investigational product (whichever is longer)
* Pregnant or lactating and breast feeding, or planning on either during the study
* Unable to comply with planned study procedures and be available for all follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who are alive and free of respiratory failure at Day 29 | Baseline through Day 29
  Proportion of subjects who are alive and free of respiratory failure at Day 29

SECONDARY OUTCOMES:
Viral load reduction | Baseline to Day 4, 15, and 29
  Log-10 viral load reduction from baseline to Day 4, Day 15, and Day 29 by nasopharyngeal RT-PCR test
Time to sustained clinical improvement | Baseline through Day 29
  Time to sustained clinical improvement defined as achieving a score of ≤2 on the Ordinal Scale for Clinical Improvement (OSCI) for a continuous period of 48h and maintained to Day 29
Proportion of subjects with clinical improvement | Baseline to Day 15 and 29
  Proportion of subjects with clinical improvement defined as ≤2 on the OSCI at Day 15 and Day 29
All-cause mortality at Day 29 | Baseline through Day 29
  All-cause mortality at Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics
Locations (1):
- Teradan Clinical Trials, Brandon, Florida, United States

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343